CLINICAL TRIAL: NCT01164124
Title: Probiotics-Supplemented Feeding in Extremely Low Birth Weight Infants
Acronym: PAS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vermont Oxford Network (Network)
Collaborators: University of Vermont (Other); St. Louis University (Other); Cardinal Glennon Children's Hospital (Unknown); Saint John Hospital & Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHRMS 08-019
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Low Birth Weight
Keywords: extremely low birth weight; probiotics; growth; nutrition; premature infants; growth in extremely low birth weight infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic supplementation (Experimental): 500 million CFU of Lactobacillus rhamnosus GG (Culturelle, Amerifit Brand Inc.) and 500 million CFU of Bifidobacterium infantis (Align, Procter & Gamble.Inc)
  Interventions: Dietary Supplement: Probiotic supplementation (Lactobacillus rhamnosus GG and Bifidobacterium infantis)
- Routine feedings (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic supplementation (Lactobacillus rhamnosus GG and Bifidobacterium infantis) — The probiotic regimen consisted of 500 million CFU of Lactobacillus rhamnosus GG (Culturelle, Amerifit Brand Inc.) and 500 million CFU of Bifidobacterium infantis (Align, Procter & Gamble.Inc)
  Arms: Probiotic supplementation
Other: Placebo — routine feedings
  Arms: Routine feedings

SUMMARY:
The overall purpose of this research is to test whether adding a supplement to the feeding of extremely low birth weight infant (infants weighing less than 2 pound 2 oz at birth) will help him/her achieve full feeding faster and achieve better weight gain.

DETAILED DESCRIPTION:
The overall purpose of this research is to test whether adding a supplement to the feeding of extremely low birth weight infant (infants weighing less than 2 pound 2 oz at birth) will help him/her achieve full feeding faster and achieve better weight gain. The study also will evaluate the benefit of that feeding supplement in decreasing the rate of infection (in the blood or in the urine) and antibiotics use in those infants.

When babies are born, the digestive system (the gastrointestinal tract) is sterile. There are no bacteria residing in their gut. When babies start feeding, it is normal for the intestine to start growing several types of bacteria. These normal (good) bacteria are thought to be helpful in keeping the intestine healthy. This is not the case in premature infants. It takes premature infants a longer time to grow bacteria in their intestines and they have fewer numbers of bacteria. In addition, the bacteria premature infants grow are not the normal one that we see in healthy infants. Instead they grow unhealthy (bad) bacteria that can potentially play a role in causing infection in the blood and urine.

Adding the normal (good) bacteria to the breast milk or infant formula might help to protect premature babies from developing blood or urine infection. In addition, adding the good bacteria might be beneficial in terms of better tolerance to milk feeding. As a result, babies may have less episodes of feeding holding and have better weight gain. Two species of bacteria, called Lactobacillus and Bifidobacteria, have been used to study this in other studies of premature babies. These two species are the most plentiful bacteria seen in the bowels of full term babies.

Participation in the study involves enrolling premature babies to receive supplement to the feeding when he/she ready to feed. Babies will be randomly assigned to receive either a bacteria (probiotic) supplement or be fed without supplement. The supplement will be added to one feeding each day. Enrolled babies will continue to get the supplement for 6-10 week. Other than the feeding supplement, being in this study will not affect care.

The main outcomes of the study will be feeding tolerance and growth. Other complications associated with prematurity, on particular infection of either the gastrointestinal tract or the blood stream will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* birth weight less than or equal to 1000 grams,
* appropriately grown for gestational age,
* age 1 to 14 days inclusive,
* intention to start enteral feeds,
* written informed consent obtained

Exclusion Criteria:

* known life-threatening congenital anomaly or condition affecting
* gastrointestinal function,
* previous NEC or gastrointestinal perforation,
* previous supplementation with probiotics
* previous enteral feedings

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Growth | 34 weeks postmenstrual age
  Percentage of infants with weight less than the 10th percentile at 34 weeks postmenstrual age.
Growth | 28 days from study entry
  Average weight gain and growth velocity during the first 28 days from initiation of feeding.
Feeding Tolerance | 28 days from study entry
  Volume of feeding per day during the first 28 days from the initiation of feeding.

SECONDARY OUTCOMES:
Antimicrobial therapy | 34 weeks post menstrual age
  Days of antimicrobial treatment until 34 weeks post menstrual age.
Complications of prematurity | until hospital discharge
  common complications of prematurity including but not limited to sepsis, necrotizing enterocolitis, and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Al-Hosni, MD, Principal Investigator — St. Louis University
Locations (3):
- United States (3):
  - St. John Hospital & Medical Center, Detroit, Michigan
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - VT Children's at Fletcher-Allen Health Care, Burlington, Vermont